CLINICAL TRIAL: NCT00687752
Title: Sonographic Assessment of Fetal Deglutition Associated With Hydramnion:Its Absence is Indicative of CNS Pathology? a Report on Two Cases.
Brief Title: Sonographic Assessment of Fetal Deglutition Associated With Hydramnion:Its Absence is Indicative of Central Nervous System (CNS) Pathology
Acronym: FD
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hippocration General Hospital (Other)
Responsible Party: assist. professor THEOHARIS TANTANASIS, 2nd department OB/GYN Hippocration General Hospital
Other Study IDs: 27052008
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2008-06-02 (Estimated); Status verified 2008-05

CONDITIONS: Hydramnios
Keywords: fetal deglutition; larynx; fetal CNS pathology; sonography; hydramnios
MeSH Terms: conditions — Polyhydramnios; Laryngeal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: hydramnios
- 2: normal

SUMMARY:
310 singleton pregnancies (22-35 weeks) enrolled into the study. We assessed sonographically the fetal larynx in an axial plane through the mandible and observed the fetal deglutition movements .

DETAILED DESCRIPTION:
310 singleton pregnancies (22-35 weeks) enrolled into the study. We assessed sonographically the fetal larynx in an axial plane through the mandible and observed the fetal deglutition movements .We encountered two cases of hydramnios were no deglutition movements could be noted. In all other cases the deglutition was normal. The motivation to conduct the current observational prospective study was to assess whether there is a link between absence of fetal deglutition and CNS pathology of the fetus. In the first case the fetus deceased at 35 weeks of gestation; obduction was declined by the parents. In the second case caesarian section at 33 weeks was carried out recently due to fetal distress. The infant is still in uncapable of swallowing and there for is under investigation at the neonatal center of our hospital.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy(22-35 weeks)

Exclusion Criteria:

* positive toxoplasmosis screening,drug and/or antidepressants addiction.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2007-05; Primary Completion 2008-04 (Estimated); Study Completion 2009-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: THEOHARIS A TANTANASIS, ASSIST PROF, Principal Investigator — 2nd dept OB/GYN ARISTOTLE UNIV. THESSALONIKI GREECE; JOHN M TZAFETTAS, PROF, Study Chair — 2nd dept OBGYN ARISTOTLE UNIV. THESSALONIKI GREECE
Locations (1):
- Hippokration General Hospital, Thessaloniki, THESSALONIKI, Greece